CLINICAL TRIAL: NCT02090595
Title: Neurofunctional Effects of Mindfulness Based Cognitive Therapy for Youth With Symptoms of Anxiety and a Familial Risk for Developing Bipolar Disorder
Brief Title: Mindfulness Based Cognitive Therapy for Youth With Anxiety at Risk for Bipolar Disorder
Acronym: Mindfulness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Melissa Delbello, MD, University of Cincinnati
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-3124
Record Dates: First submitted 2014-03-13; First posted 2014-03-18 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2015-05

CONDITIONS: Anxiety; Bipolar Disorder
Keywords: bipolar disorder; anxiety; mindfulness; high risk; cognitive behavioral
MeSH Terms: conditions — Anxiety Disorders; Bipolar Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MBCT-C (Experimental): Mindfulness-Based Cognitive Therapy for Anxious Children (MBCT-C) is a 12-week manualized group therapy program for children with anxiety disorders. The program involves teaching children to pay attention to anxiety-related thoughts, emotions, and physical sensations with openness and non-judgment.
  Interventions: Behavioral: MBCT-C
- Waitlist Control (Other): Education and Therapy
  Interventions: Behavioral: Waitlist Control

INTERVENTIONS:
Behavioral: MBCT-C — A 12 week group therapy program for children with anxiety disorders. This involves teaching the children the pay attention to anxiety related cues with openness and non-judgment. Group leaders begin each session with: sitting meditation, review of the previous session and home practices, teaching a new mindfulness exercise, reading a group poem or story, distributing handouts, etc. There will be a new theme each week.
  Arms: MBCT-C
Behavioral: Waitlist Control — Waitlist Control (WC) will be the comparison condition. Some of the children in the study will initially participate in a 12 week WC prior to their participation in the MBCT-C. At each visit during the waitlist control period, participants and their families will receive materials about mood and anxiety disorders in youth, bipolar disorders, familial risk for bipolar disorder and treatment strategies for anxiety and depression in youth.
  Arms: Waitlist Control

SUMMARY:
Children who have parents with bipolar disorder are at risk for developing anxiety disorders.

DETAILED DESCRIPTION:
Children who have parents with bipolar disorder are at risk for developing anxiety disorders. Typical treatments for anxiety in children are SSRI antidepressants. However, these medications may accelerate the onset of mania or hypomania in children with a family history of bipolar disorder or cause suicidal thinking in children. Studies trying alternative treatments to anxiety and possible bipolar disorder in children are needed, to establish other methods for treating childhood mental health. These studies can also help with early intervention and possible future prevention strategies for bipolar disorder. This study involves treating anxious children with Mindfulness Based Cognitive Therapy. They will have 12 weeks of mindfulness therapy in a group with other children where they will be led by a trained group leader, how to pay attention to anxiety cues and react differently.

ELIGIBILITY:
Inclusion Criteria:

* 10-17 years old
* At least one parent with bipolar disorder
* Meets clinical criteria for a specific anxiety disorder
* PARS -5 item scale score > 10 at screening and baseline of initial study phase
* Fluent in English;
* Provision of written informed consent/assent
* Agrees to participate in 75% of sessions

Exclusion Criteria:

CANNOT Have any of the Following:

* Documented diagnosis of mental retardation or IQ <70
* Previous participation in mindfulness-based treatment
* Substance use disorder within last 3 months
* Judged clinically to be suicide risk
* Concurrent treatment with psychotropic medication (certain exceptions apply, ask for details)
* Psychotherapy initiated within 2 months prior to screening or plan to initiate psychotherapy during study participation
* Any lifetime diagnosis of bipolar disorder, cyclothymia, schizophrenia, or other psychotic disorder
* Any symptom that requires admission to an inpatient psychiatric unit
* Anxiety symptoms resulting from acute medical illness or acute intoxication or withdrawal from drugs or alcohol

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2013-07; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
The Pediatric Anxiety Rating Scale | 12 weeks
  Change from baseline to endpoint in the Pediatric Anxiety Rating Scale (PARS) score. The PARS is a rating scale (a form that a clinician fills out) to determine the severity of anxiety in children.

SECONDARY OUTCOMES:
Change in other Anxiety | 12 weeks
  The STAI-C is a rating scale that will determine the severity of state and trait related anxiety symptoms over time. State anxiety will be assessed at each visit. Trait anxiety will be assessed at Screening.Baseline and Week 12.
Mood | 12 weeks
  The Children's Depression Rating Scale-Revised (CDRS) will measure symptoms of depression and the Young Mania Rating Scale (YMRS) will measure symptoms of mania.
Behavioral | 12 weeks
  The Child Behavior Checklist (CBCL) is a rating scale to examine a child's behavior.
Quality of Life | 12 weeks
  The Children's Global Assessment Score (CGAS) and the Children Health Questionnaire (CHQ) are rating scales that will determine a child's quality of life.

OTHER OUTCOMES:
Potential Mediators | 12 weeks
  Exploration of whether or not measures of mindfulness, emotional deregulation and attention will serve as potential mediators. The hypothesis that increased mindfulness, emotional regulation, and attention will mediate treatment-related improvements in anxiety, mood and behavior and QOL will be evaluated using structural equation models.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa DelBello, MD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided